CLINICAL TRIAL: NCT05699733
Title: Influences of Mechanical Traction Using Different Forces on Knee Joint Space, Range of Motion, and Hamstring Flexibility in Asymptomatic Subjects: Preliminary Study
Brief Title: Mechanical Traction Force and Knee Joint Space
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, assistant professor, University of Hail
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-2022-403
Record Dates: First submitted 2022-11-08; First posted 2023-01-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Knee Arthritis

STUDY DESIGN:
Intervention Model Description: the recruited sample will be subjected to 3 treatment conditions according to the traction force used. pre-post comparisons and between conditions comparisons will be conducted
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechanical traction force 30% of body weight (Experimental): will receive continuous mechanical traction from semi flexed knee, for 30 minutes using 30% of the body weight as a traction force
  Interventions: Device: mechanical traction for knee joint
- Mechanical traction force 20% of body weight (Experimental): will receive continuous mechanical traction from semi flexed knee, for 30 minutes using 20% of the body weight as a traction force
  Interventions: Device: mechanical traction for knee joint
- Mechanical traction force 10% of body weight (Experimental): will receive continuous mechanical traction from semi flexed knee, for 30 minutes using 10 % of the body weight as a traction force
  Interventions: Device: mechanical traction for knee joint

INTERVENTIONS:
Device: mechanical traction for knee joint — All participants will receive a single session per condition. This session will consist of continuous mechanical knee traction for 30 minutes while the participant assumes a supine position with the treated limb in semiflexion (30° of flexion). the treated limb will be supported using the traction bed's table that is used for this purpose. The knee position angle will be measured by a standard goniometer. Pelvis and thigh straps will be used to fix the body and prevent slippage during the application of the traction force. A customized leg cuff will be placed around the lower leg (above the ankle joint), and a traction rope will be extending horizontally from the cuff to the traction device. 48 hours of washing out will separate the sessions of different conditions

SUMMARY:
the purposes of this crossover study are to Purpose

1. To determine the most effective traction force for knee joint that can be used in the treatment of patients with KOA.
2. To determine the influence of knee joint traction on ROM ok knee joint flexion and extension
3. To determine the influence of knee joint traction on the flexibility of hamstring muscles

DETAILED DESCRIPTION:
this study is a pilot study design aiming to determine the most effective mechanical traction force used for knee joint treatment. this effectiveness was assessed in favor of the separation of the joint surfaces in cm in addition to the hamstring flexibility measured in cm and active knee flexion range of motion.

according to previous literature, there is no consensus regarding the most appropriate traction force that can produce statistical and clinically meaningful differences so we started this pilot study.

the results of this study will be used to conduct a larger-scale study using the most appropriate traction force on patients having knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subject
2. males or females
3. No previous surgery in lower limbs

Exclusion Criteria:

1. Diseased knee joint
2. Knee osteoarthritis
3. Any musculoskeletal problem in the lower extremities
4. Varicose veins
5. Pregnancy

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
knee joint space | immediate (after first session)
  the distance in millimeters will be measured between the articilar acriliges of femur and tibia in non-weight bearing position from the medial and lateral aspects of the knee joint using ultrasonography device designed to assess musculoskeletal conditions
knee joint space | short term (30 minutes after the first session)
  the distance in millimeters will be measured between the articilar acriliges of femur and tibia in non-weight bearing position from the medial and lateral aspects of the knee joint using ultrasonography device designed to assess musculoskeletal conditions

SECONDARY OUTCOMES:
hamstrings flexibility | immediate (after first session)
  using the Sit and reach test: The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back. it is also a field test which is easy to administer in a community setting with a large scale of population size
hamstrings flexibility | short term (30 minutes after the first session)
  using the Sit and reach test: The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back. it is also a field test which is easy to administer in a community setting with a large scale of population size
knee active range of motion | immediate (after first session)
  Bubble inclinometer will be used to assess the active knee joint flexion range. Participant will assume supine position and after proper placement of the goniometer, she will be asked to bend her knee and hip joints as much as possible
knee active range of motion | short term (30 minutes after the first session)
  Bubble inclinometer will be used to assess the active knee joint flexion range. Participant will assume supine position and after proper placement of the goniometer, she will be asked to bend her knee and hip joints as much as possible

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hail, Hail, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
it will available upon request from the principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year